CLINICAL TRIAL: NCT00432744
Title: Phase 3 Trial of Coenzyme Q10 in Mitochondrial Disease
Brief Title: Phase III Trial of Coenzyme Q10 in Mitochondrial Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01FD003032-01A1 (FDA); R01FD003032-01A1 (FDA)
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Mitochondrial Diseases
Keywords: mitochondrial diseases; respiratory chain complex I deficiencies; respiratory chain complex II deficiencies; respiratory chain complex III deficiencies; respiratory chain complex IV deficiencies; mutations of a gene coding for a respiratory chain component
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CoenzymeQ10 (Active Comparator): CoenzymeQ10: patients will be randomized to receive CoenzymeQ10 in either Period #1 (Months 0-6) or Period #2 (Months 7-12).
  Interventions: Drug: CoenzymeQ10
- Placebo (Placebo Comparator): Placebo: patients will be randomized to receive placebo either ion Period #1 (months 1-6) or Period #2 (months 7-12).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CoenzymeQ10 — CoenzymeQ10 will be given in 10 mg/kg daily up to 400 mg. Then a draw of CoQ10 troughs every three months will be performed.
  Arms: CoenzymeQ10
Drug: Placebo — Placebo will be given in 10 mg/kg daily up to 400 mg. Then a draw of placebo troughs every three months will be performed. This treatment group will be treated as the active group.
  Arms: Placebo

SUMMARY:
To show that oral CoQ10 is a safe and effective treatment for children with inborn errors of mitochondrial energy metabolism due to defects in specific respiratory chain (RC) complexes or mitochondrial DNA (mtDNA) mutations, and that this beneficial action is reflected in improved motor and neurobehavioral function.

DETAILED DESCRIPTION:
In many patients mitochondrial disease leads to progressive nerve and muscle damage that may be associated with problems with thinking, talking, remembering, walking or balancing. Sometimes it may also cause abnormal build up in the blood and spinal fluid of a substance called lactic acid. This problem makes the blood and spinal fluid too acid, which can be life-threatening. There is no known specific or effective treatment for mitochondrial diseases. Sometimes certain diets can improve the condition but seldom prevent the nerve or muscle damage or reduce the chance of developing life-threatening acidity of the blood.

CoQ10 is not approved by the Food and Drug Administration (FDA) for the treatment of mitochondrial diseases. It is an investigational drug that we believe may help people with certain mitochondrial diseases, like the one you have, both in terms of reducing the acidity of your blood and preventing or decreasing nerve and muscle damage. Our belief is based on previous studies that have been conducted in children with mitochondrial diseases of various types. Therefore, a 12 month study has been designed to determine the safety and benefit of taking CoQ10 every day. This will be done by comparing the subjects response to taking CoQ10 for 6 months to taking a placebo for 6 months. A placebo looks, smells, and tastes like the drug being tested (in this case, CoQ10) but has no effect. Placebo studies such as this one are very common in evaluating investigational drugs for any disease and are usually required by the FDA before a drug can be approved.

CoQ10 or placebo will be given as a liquid once per day in the evening, by mouth or feeding tube. The CoQ10 dose will be 10 mg/kg with a maximum dose of 400 mg a day. Neither the subject nor the health care givers will know exactly when subjects are receiving CoQ10 or when subjects are receiving the placebo. However, subjects will receive CoQ10 for at least 6 months. At each visit the subject will be given a seven month supply of CoQ10, nutritional cocktail, and multivitamins to take home and they will be asked to bring back any unused medications at the next visit. At each visit subjects will be given a medication diary to record the time and date that they take the medications that will be provided. This diary should be returned to the study coordinator at the subject's scheduled visit. During the 12 month period that subjects are on the study, they will be expected to stop taking all medications and other supplements except for those provided by the study and those that the study doctor determines are medically needed. Except in the case of an emergency, the subject must contact the study doctor before taking any new medications or supplements. In the case of an emergency, subjects are required to inform the study doctor of the emergency and treatments as soon as possible.

Subjects will be hospitalized on the General Clinical Research Center (GCRC) ward of Shands Hospital for 2-4 days every three to six months. A parent or legal guardian will be expected to stay with the subject. During that hospitalization, physical and intellectual development will be measured by standard tests. The GCRC dietician will ask questions about current diet at each visit and record answers. A general medical history and physical examination (including gross motor function and/or strength tests) will be performed during each visit as well as a six minute walking test. While enrolled in this study, a special "nutritional cocktail" and a Centrum-like multivitamin supplement will be provided for subjects to take daily. The nutritional cocktail has vitamin C, up to 10 mg/kg/day (max. 400 mg/day), riboflavin, up to 2.5 mg/kg/day (max. 100 mg/day), thiamine, up to 2.5 mg/kg/day (100 mg/day), carnitine, up to 10 mg/kg/day (max. 400 mg/day). The nutritive cocktail is in capsule form and the number of capsules that the subject will take will be based on body weight (for every 4 kg. of body weight subjects will receive 1 capsule daily). Each capsule contains: Vitamin C 40 mg, Riboflavin 10 mg, thiamine 10 mg and carnitine 40 mg. The maximum amount of capsules that will be given daily to anyone in this study is 10 capsules daily. A parent or legal guardian will be asked to complete each of eight questionnaires regarding behavioral and developmental, quality of life (5), and sleep. The behavioral and developmental, four of the quality of life (QOL) questionnaires, and the sleep questionnaire should be completed at the 0, 6 and 12 month visits. One of the QOL questionnaires (46 questions) will need to be completed monthly and mailed back to the study center after completion (self-addressed, stamped envelopes will be provided by the study and given to you by the coordinator). We expect that it will take up to 20 minutes to complete the monthly QOL questionnaire and up to 3 hours at the 0, 6 and 12 month visit to complete the rest of the questionnaires.

About 15-20 ml. of blood (3-4 teaspoons) will be obtained during each hospitalization. A urine sample will also be collected during each hospital visit. In females of child-bearing age, urine will also be collected and tested for the presence of HCG (a hormone that determines pregnancy). Within 24 hours of blood and urine collection test results will be assessed by the study physician.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 m - 17 y
* Biochemical proof of a deficiency of complex I, III or IV of the RC or a molecular genetic proof of a mutation in mtDNA, or an nDNA mutation in a gene known to be associated with dysfunction of the electron transport chain (e.g., SURF1)
* Willingness to stop all other medication regimens and supplements other than what the Steering and Planning Committee deems medically necessary

Exclusion Criteria:

* A genetic mitochondrial disease other than those stipulated under inclusion criteria
* Intractable epilepsy, defined as grand mal seizures occurring with a frequency > 4/month, despite treatment with conventional antiepileptic drugs
* Primary, defined organic acidurias other than lactic acidosis (e.g., propionic aciduria
* Primary disorders of amino acid metabolism
* Primary disorders of fatty acid oxidation
* Secondary lactic acidosis due to impaired oxygenation or circulation (e.g., due to severe cardiomyopathy or congenital heart defects)
* Severe anemia, defined as a hematocrit <30%
* Malabsorption syndromes associated with D-lactic acidosis
* Renal insufficiency, defined as (1) a requirement for chronic dialysis or (2) serum creatinine ≥ 1.2 mg/dl or creatinine clearance <60 ml/min
* Primary hepatic disease unrelated to mitochondrial disease
* Allergy to CoQ10 or placebo ingredients
* Pregnancy

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2007-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S. Kerr, MD, PhD, Principal Investigator — Case Western Reserve University; Ton J deGrauw, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Annette S. Feigenbaum, MD, Principal Investigator — SickKids, Toronto, Canada/University of Toronto
Locations (3):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hanna MG, Nelson IP. Genetics and molecular pathogenesis of mitochondrial respiratory chain diseases. Cell Mol Life Sci. 1999 May;55(5):691-706. doi: 10.1007/s000180050327. PMID 10379358
- [Background] Kerr DS. Treatment of congenital lactic acidosis: a review. Intern Pediatr, 1995;10:75-81.
- [Background] Abe K, Fujimura H, Nishikawa Y, Yorifuji S, Mezaki T, Hirono N, Nishitani N, Kameyama M. Marked reduction in CSF lactate and pyruvate levels after CoQ therapy in a patient with mitochondrial myopathy, encephalopathy, lactic acidosis and stroke-like episodes (MELAS). Acta Neurol Scand. 1991 Jun;83(6):356-9. doi: 10.1111/j.1600-0404.1991.tb03962.x. PMID 1887756
- [Background] Ogasahara S, Nishikawa Y, Yorifuji S, Soga F, Nakamura Y, Takahashi M, Hashimoto S, Kono N, Tarui S. Treatment of Kearns-Sayre syndrome with coenzyme Q10. Neurology. 1986 Jan;36(1):45-53. doi: 10.1212/wnl.36.1.45. PMID 3941783
- [Background] Gold R, Seibel P, Reinelt G, Schindler R, Landwehr P, Beck A, Reichmann H. Phosphorus magnetic resonance spectroscopy in the evaluation of mitochondrial myopathies: results of a 6-month therapy study with coenzyme Q. Eur Neurol. 1996;36(4):191-6. doi: 10.1159/000117246. PMID 8814419
- [Background] Matthews PM, Ford B, Dandurand RJ, Eidelman DH, O'Connor D, Sherwin A, Karpati G, Andermann F, Arnold DL. Coenzyme Q10 with multiple vitamins is generally ineffective in treatment of mitochondrial disease. Neurology. 1993 May;43(5):884-90. doi: 10.1212/wnl.43.5.884. PMID 8492942
- [Background] Bresolin N, Doriguzzi C, Ponzetto C, Angelini C, Moroni I, Castelli E, Cossutta E, Binda A, Gallanti A, Gabellini S, et al. Ubidecarenone in the treatment of mitochondrial myopathies: a multi-center double-blind trial. J Neurol Sci. 1990 Dec;100(1-2):70-8. doi: 10.1016/0022-510x(90)90015-f. PMID 2089142
- [Background] Shults CW, Oakes D, Kieburtz K, Beal MF, Haas R, Plumb S, Juncos JL, Nutt J, Shoulson I, Carter J, Kompoliti K, Perlmutter JS, Reich S, Stern M, Watts RL, Kurlan R, Molho E, Harrison M, Lew M; Parkinson Study Group. Effects of coenzyme Q10 in early Parkinson disease: evidence of slowing of the functional decline. Arch Neurol. 2002 Oct;59(10):1541-50. doi: 10.1001/archneur.59.10.1541. PMID 12374491
- [Background] Ogasahara S, Engel AG, Frens D, Mack D. Muscle coenzyme Q deficiency in familial mitochondrial encephalomyopathy. Proc Natl Acad Sci U S A. 1989 Apr;86(7):2379-82. doi: 10.1073/pnas.86.7.2379. PMID 2928337
- [Background] Musumeci O, Naini A, Slonim AE, Skavin N, Hadjigeorgiou GL, Krawiecki N, Weissman BM, Tsao CY, Mendell JR, Shanske S, De Vivo DC, Hirano M, DiMauro S. Familial cerebellar ataxia with muscle coenzyme Q10 deficiency. Neurology. 2001 Apr 10;56(7):849-55. doi: 10.1212/wnl.56.7.849. PMID 11294920
- [Background] Lamperti C, Naini A, Hirano M, De Vivo DC, Bertini E, Servidei S, Valeriani M, Lynch D, Banwell B, Berg M, Dubrovsky T, Chiriboga C, Angelini C, Pegoraro E, DiMauro S. Cerebellar ataxia and coenzyme Q10 deficiency. Neurology. 2003 Apr 8;60(7):1206-8. doi: 10.1212/01.wnl.0000055089.39373.fc. PMID 12682339
- [Background] Rahman S, Hargreaves I, Clayton P, Heales S. Neonatal presentation of coenzyme Q10 deficiency. J Pediatr. 2001 Sep;139(3):456-8. doi: 10.1067/mpd.2001.117575. PMID 11562630
- [Background] Argov Z, Bank WJ, Maris J, Eleff S, Kennaway NG, Olson RE, Chance B. Treatment of mitochondrial myopathy due to complex III deficiency with vitamins K3 and C: A 31P-NMR follow-up study. Ann Neurol. 1986 Jun;19(6):598-602. doi: 10.1002/ana.410190615. PMID 3014998
- [Background] Geromel V, Darin N, Chretien D, Benit P, DeLonlay P, Rotig A, Munnich A, Rustin P. Coenzyme Q(10) and idebenone in the therapy of respiratory chain diseases: rationale and comparative benefits. Mol Genet Metab. 2002 Sep-Oct;77(1-2):21-30. doi: 10.1016/s1096-7192(02)00145-2. PMID 12359126
- [Background] Beal MF. Mitochondria, oxidative damage, and inflammation in Parkinson's disease. Ann N Y Acad Sci. 2003 Jun;991:120-31. doi: 10.1111/j.1749-6632.2003.tb07470.x. PMID 12846981
- [Background] Turunen M, Olsson J, Dallner G. Metabolism and function of coenzyme Q. Biochim Biophys Acta. 2004 Jan 28;1660(1-2):171-99. doi: 10.1016/j.bbamem.2003.11.012. PMID 14757233
- [Background] Miles MV, Horn PS, Tang PH, Morrison JA, Miles L, DeGrauw T, Pesce AJ. Age-related changes in plasma coenzyme Q10 concentrations and redox state in apparently healthy children and adults. Clin Chim Acta. 2004 Sep;347(1-2):139-44. doi: 10.1016/j.cccn.2004.04.003. PMID 15313151
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Cerveri I, Fanfulla F, Zoia MC, Manni R, Tartara A. Sleep disorders in neuromuscular diseases. Monaldi Arch Chest Dis. 1993 Aug;48(4):318-21. PMID 8257973
- [Background] Johnston K, Newth CJ, Sheu KF, Patel MS, Heldt GP, Schmidt KA, Packman S. Central hypoventilation syndrome in pyruvate dehydrogenase complex deficiency. Pediatrics. 1984 Dec;74(6):1034-40. PMID 6438601
- [Background] Kotagal S, Archer CR, Walsh JK, Gomez C. Hypersomnia, bithalamic lesions, and altered sleep architecture in Kearns-Sayre syndrome. Neurology. 1985 Apr;35(4):574-7. doi: 10.1212/wnl.35.4.574. PMID 3982647
- [Background] Pronicka E, Piekutowska-Abramczuk DH, Popowska E, Pronicki M, Karczmarewicz E, Sykut-Cegielska Y, Taybert J. Compulsory hyperventilation and hypocapnia of patients with Leigh syndrome associated with SURF1 gene mutations as a cause of low serum bicarbonates. J Inherit Metab Dis. 2001 Dec;24(7):707-14. doi: 10.1023/a:1012937204315. PMID 11804207
- [Background] Sakaue S, Ohmuro J, Mishina T, Miyazaki H, Yamaguchi E, Nishimura M, Fujita M, Nagashima K, Tagami S, Kawakami Y. A case of diabetes, deafness, cardiomyopathy, and central sleep apnea: novel mitochondrial DNA polymorphisms. Tohoku J Exp Med. 2002 Mar;196(3):203-11. doi: 10.1620/tjem.196.203. PMID 12002277
- [Background] Spranger M, Schwab S, Wiebel M, Becker CM. [Adult Leigh syndrome. A rare differential diagnosis of central respiratory insufficiency]. Nervenarzt. 1995 Feb;66(2):144-9. German. PMID 7715756
- [Background] Yasaki E, Saito Y, Nakano K, Katsumori H, Hayashi K, Nishikawa T, Osawa M. Characteristics of breathing abnormality in Leigh and its overlap syndromes. Neuropediatrics. 2001 Dec;32(6):299-306. doi: 10.1055/s-2001-20405. PMID 11870585
- [Background] Sembrano E, Barthlen GM, Wallace S, Lamm C. Polysomnographic findings in a patient with the mitochondrial encephalomyopathy NARP. Neurology. 1997 Dec;49(6):1714-7. doi: 10.1212/wnl.49.6.1714. PMID 9409376
- See also: University of Florida Clinical Research Center, Clinical and Translational Science Institute — https://www.ctsi.ufl.edu/research/clinical-research-units-n-z/uf-clinical-research-center/
- See also: Describes the 23 item Pediatric Quality of Life — http://www.pedsql.org/about_pedsql.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo First: Patients will be randomized to receive Placebo in Period #1 (Months 0-6) and CoenzymeQ10 given in Period #2( Months 7-12.)
  Placebo: Placebo will be given in 10 mg/kg daily up to 400 mg. Then a draw of placebo troughs every three months will be performed. This treatment group will be treated as the active group.
  CoenzymeQ10: CoenzymeQ10 will be given in 10 mg/kg daily up to 400 mg. Then a draw of CoQ10 troughs every three months will be performed.
- CoenzymeQ10 Frist: Patients will be randomized to receive CoenzymeQ10 in Period #1 (Months 0-6) and Placebo given in Period #2( Months 7-12.)
  CoenzymeQ10: CoenzymeQ10 will be given in 10 mg/kg daily up to 400 mg. Then a draw of CoQ10 troughs every three months will be performed.
  Placebo: Placebo will be given in 10 mg/kg daily up to 400 mg. Then a draw of placebo troughs every three months will be performed. This treatment group will be treated as the active group.
Period: Months 0-6
Arm/Group | Placebo First | CoenzymeQ10 Frist
Started | 12 | 12
Completed | 7 | 8 (One patient in period 1 "other reason" for loss became too disabled to complete the 6 month test.)
Not Completed | 5 | 4
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Too disabled to score | 1 | 0
Period: Months 7 - 12
Arm/Group | Placebo First | CoenzymeQ10 Frist
Started | 7 | 8
Completed | 6 | 7
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Too disabled to score | 0 | 1

BASELINE CHARACTERISTICS:
Population: This is the set of subjects that met all eligibility requirements
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo First | CoenzymeQ10 Frist | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (6.3) | 7.5 (4.5) | 8.3 (5.4)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19
  Canada | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: McMaster Gross Motor Function (GMFM 88)
Description: The McMaster Gross Motor Function is a validated scale ranging from 0 to 100 (the higher the better). Since there was the possibility of a subject becoming totally disabled our FDA peer reviewed design called for its use as follows: If the subject completed both periods, the score was calculated as the difference in scores between the end of Period 2 (at 12 months) minus that at the end of Period 1 (6 months). If a subject became totally disabled, this difference was considered as plus infinity if it occurred in period 1 (Penalizes period 1), and minus infinity if it occurred in Period 2 (Penalizes period 2). The two treatments were compared via the Wilcoxon test, and the effect size was estimated using Kendall's Tau-B. This is interpreted in a similar manner to correlation with positive values favoring COQenzyme10 and negative values favoring placebo. One of the links in this report is to the the GMFM scale and how it is scored. A link to the instrument is included.
Time Frame: Taken at 6 and 12 Months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First | CoenzymeQ10 Frist
Number analyzed (Participants) | 6 | 8
units on a scale | -0.002 [-0.47 to 1.36] | -0.12 [-2.75 to 1.75]
Statistical Analysis 1: Comparison: Placebo First vs CoenzymeQ10 Frist; Study intended to accrue 40 subjects, but only obtained 14 evaluable on this endpoint; Test type: Superiority or Other; p = 0.95, Wilcoxon (Mann-Whitney) — Two-sided Test; Kendall's Tau B = .015, 95% CI 2-sided [-0.44 to 0.48], Standard Error of Mean 0.23 — Positive value of Tau-B would favor CoQ

2. Primary Outcome: Pediatric Quality of Life Scale
Description: The Pediatric Quality of Life Scale is a validated scale ranging from 0 to 100 (the higher the better). Since there was the possibility of a subject becoming totally disabled our FDA peer reviewed design called for its use as follows: If the subject completed both periods, the score was calculated as the difference in scores between the end of Period 2 (at 12 months) minus that at the end of Period 1 (6 months). If a subject became totally disabled, this difference was considered as plus infinity if it occurred in period 1 (Penalizes period 1), and minus infinity if it occurred in Period 2 (Penalizes period 2). The two treatments were compared via the Wilcoxon test, and the effect size was estimated using Kendall's Tau-B. This is interpreted in a similar manner to correlation with positive values favoring COQenzyme10 and negative values favoring placebo. Goggle "pedsQL and Mapi" to browse the copyrighted manual. A link to the instrument is included.
Time Frame: At 6 and 12 Months
Population: 7 subjects in each group were evaluable for this endpoint. The two subjects who became disabled are evaluable. One subject did not have period 2 Quality of Life data and is excluded.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Placebo First | CoenzymeQ10 Frist
Number analyzed (Participants) | 7 | 7
units on a scale | -1.1 [-4.3 to 7.1] | -11.9 [-43.5 to 4.3]
Statistical Analysis 1: Comparison: Placebo First vs CoenzymeQ10 Frist; Study intended to accrue 40 subjects, but only obtained 14 evaluable on this endpoint; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney); Kendall's Tau B = 0.30, 95% CI 2-sided [-0.12 to 0.72], Standard Error of Mean 0.21 — A positive value would favor CoQ

3. Primary Outcome: Non-parametric Hotelling T-square Bivariate Analysis of GMGF 88 and OPeds QOL.
Description: This is a multivariate analysis of the first two outcomes: Period 2 minus Period 1 GMFM88 and Peds Quality of Life, analyzed as follows: First, to be in the analysis, subjects must contribute at least one of these endpoints. Second, if the subject became totally disabled during period 1, the difference was defined as + infinity, (highest possible evidence favoring period 2), and if the subject became totally disabled in period 2, the subject was scored as - infinity (highest possible evidence favoring period 1). Period 2 minus period 1 differences were ranked form low to high with missing values scores at the mid-rank. The Hotelling T-square was computed on these ranks and the P-value was obtained from 100,000 rerandomizations as the fraction of rerandomizations with T-sq at least as large as that observed.
Time Frame: end of 12 month minus end of 6 month difference.
Population: Subjects contributes at least one difference (either GMFM or Peds QOL). Thirteen contributed both and one each was missing GMFM or Peds QOL.
Measure: Number; unit: participants
Arm/Group | Placebo First | CoenzymeQ10 Frist
Number analyzed (Participants) | 7 | 8
participants | 7 | 8
Statistical Analysis 1: Comparison: Placebo First; The actual study was powered to have 40 participants but only 24 participated and of these only 15 had outcome data; Test type: Superiority or Other; p = 0.42, Non-parametric Hotelling T-square — The Hotelling T-sq=1.74 and 42% of the rerandomizations to groups of 7 and 8 had Hotelling T-sq of at least 1.74. This is the standard method for permutation tests. The large sample null is chi-sq with 2 df, which has a mean=2

ADVERSE EVENTS:
Time Frame: AE's were collected from 10/2007 to 4/2012.
Groups:
- CoenzymeQ10: CoenzymeQ10: CoenzymeQ10 will be given in 10 mg/kg daily up to 400 mg. Then a draw of CoQ10 troughs every three months will be performed. (Either in Period 1 or Period 2)
- Placebo: Placebo: Placebo will be given in 10 mg/kg daily up to 400 mg. Then a draw of placebo troughs every three months will be performed. This treatment group will be treated as the active group. (Either in Period 1 or Period 2)
Arm/Group | CoenzymeQ10 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/20
Other Adverse Events (participants affected / at risk) | 10/19 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoenzymeQ10 (N=19) | Placebo (N=20)
Hospitalization for lumbar vertebrae fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Subject was involved in an accident in which two (2) lumber vertebrae were fractured
Altered Mental State (Nervous system disorders) | 0 (0) | 1 (1) — Not related to the study
Hospitalization for seizure activity (Nervous system disorders) | 1 (1) | 0 (0) — Subject with MELAS; not related to study
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CoenzymeQ10 (N=19) | Placebo (N=20)
Decreased White Blood Count (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Low ANC Levels (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nose Bleed (General disorders) | 0 (0) | 1 (1)
Elevated Liver Enzymes (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 1 (1) | 1 (1)
GI Issues (Gastrointestinal disorders) | 2 (2) | 5 (5)
Fatigue (General disorders) | 1 (1) | 0 (0)
Neuromusclar Changes (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Mental Status Change (Nervous system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
GTube Infection (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial intended to accrual 40 subjects, but accrual was below expectations and the granting agency turned down a request for extended accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No